CLINICAL TRIAL: NCT00435370
Title: Tropisetron With Risperidone for Schizophrenia
Brief Title: Effectiveness of Tropisetron Plus Risperidone for Improving Cognitive and Perceptual Disturbances in Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Thomas R. Kosten, MD, Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: U01MH079639 (NIH); U01MH079639 (NIH)
Record Dates: First submitted 2007-02-13; First posted 2007-02-14 (Estimated); Results first posted 2014-09-08 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-02

CONDITIONS: Smoking Cessation; Schizophrenia
MeSH Terms: conditions — Smoking Cessation; Schizophrenia | interventions — Tropisetron; Risperidone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tropisetron (Experimental): Tropisetron (10mg/day) + risperidone(6mg/day)
  Interventions: Drug: Tropisetron; Drug: Risperidone
- Placebo (Placebo Comparator): Placebo + risperidone (6mg/day)
  Interventions: Drug: Placebo; Drug: Risperidone

INTERVENTIONS:
Drug: Tropisetron — 10 mg/day
  Other Names: Navoban
  Arms: Tropisetron
Drug: Placebo — placebo
  Arms: Placebo
Drug: Risperidone — 6mg/day
  Other Names: Risperdal, Ridal, Rispolept

SUMMARY:
This study will determine the effectiveness of tropisetron plus risperidone in improving cognitive symptoms in Chinese people with schizophrenia.

DETAILED DESCRIPTION:
Schizophrenia is a chronic and disabling brain disorder. People with schizophrenia may experience hallucinations, delusions, disordered thinking, movement disorders, social withdrawal, and cognitive deficits. In considering the high rate of cigarette smoking among people with schizophrenia, it is also likely that they smoke. People with schizophrenia who smoke tend to experience improved cognition, and tobacco withdrawal has been associated with deterioration of cognition. This suggests that nicotine may improve cognitive deficits or medication side effects in people with schizophrenia.

Auditory sensory gating, a neural mechanism thought to reflect sensory information processing and affect cognition, is diminished in people with schizophrenia. Auditory sensory gating has been associated with the 7 nicotinic acetylcholine receptor, a brain receptor that is important for cognition and can be activated by nicotine. Activation of this receptor using an agonist medication, such as tropisetron, may produce the same positive effect that nicotine has on cognition. This study will determine the effectiveness of using tropisetron as supplemental therapy to the atypical neuroleptic risperidone in people with schizophrenia.

Participants in this 12-week double blind study will be randomly assigned to receive either tropisetron or placebo. All participants will also follow a 6-mg risperidone regimen. Study visits will occur every 2 weeks throughout the study and final outcome assessments will include cognitive functioning and treatment safety and effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Currently resides in Beijing, China
* Diagnosis of schizophrenia or schizophreniform disorder
* Duration of symptoms is no longer than 60 months
* No history of treatment with antipsychotic medication or, if previously treated, a total lifetime usage of less than 14 days
* Current psychotic symptoms are of moderate severity or greater as measured by one of the five psychotic items in the Brief Psychiatric Rating Scale (BPRS)

Exclusion Criteria:

* Diagnostic and Statistical Manual of Mental Disorders(DSM)-IV Axis I diagnosis other than schizophrenia or schizophreniform psychosis
* Documented disease of the central nervous system that might interfere with the trial assessments (e.g., stroke, tumor, Parkinson's disease, Huntington's disease, seizure disorder, history of brain trauma resulting in significant impairment, chronic infection)
* Acute, unstable, and/or significant and untreated medical illness (e.g., infection, unstable diabetes, uncontrolled hypertension)
* A clinically significant echocardiogram (ECG) abnormality in the opinion of the investigator
* Pregnant or breastfeeding
* Use of prohibited concomitant therapy
* History of severe allergy or hypersensitivity
* Dependence on alcohol or illegal drugs
* Use of any of the following medications during the trial: antipsychotic medications other than risperidone; psychostimulants; or antidepressants

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 179 (Actual)
Dates: Start 2006-11; Primary Completion 2011-02 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kosten, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- Baylor College of Medicine - Michael E. DeBakey VA Medical Center, Houston, Texas, United States
- Beijing Hui-Long Guan Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang M, Liu L, Cui H, Deng C, Xiong W, Zhao G, Du S, Kosten TR, Chen H, Li Z, Zhang X. Dynamic functional thalamocortical dysconnectivity in schizophrenia correlates to antipsychotics response. Schizophrenia (Heidelb). 2023 Jul 4;9(1):40. doi: 10.1038/s41537-023-00371-y. PMID 37402747
- [Derived] Zhang XY, Liu L, Liu S, Hong X, Chen DC, Xiu MH, Yang FD, Zhang Z, Zhang X, Kosten TA, Kosten TR. Short-term tropisetron treatment and cognitive and P50 auditory gating deficits in schizophrenia. Am J Psychiatry. 2012 Sep;169(9):974-81. doi: 10.1176/appi.ajp.2012.11081289. PMID 22952075

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period began in May 2006 and ended in April 2011. Participants were approached for participation in this study after being hospitalized for at least 2 weeks if they were schizophrenic and capable of providing written informed consent.
Pre-assignment Details: After signing informed consent for participation in the study, subjects were interviewed by study doctor and all medical and psychiatric data were reviewed prior to admitting the subject and beginning medication.
Period: Overall Study
Arm/Group | Tropisetron | Placebo
Started | 90 | 89 (The recruitment restarted in August, 2010.)
Completed | 68 | 69 (The entire recruitment has been completed in December, 2011.)
Not Completed | 22 | 20
Not completed — Adverse Event | 8 | 8
Not completed — Withdrawal by Subject | 10 | 10
Not completed — Antipsychotic medication changed | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tropisetron | Placebo | Total
Number analyzed (Participants) | 90 | 89 | 179
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 90 | 89 | 179
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.8 (9.2) | 28.3 (9.9) | 28.6 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 50 | 102
  Male | 38 | 39 | 77
Region of Enrollment [Number; unit: participants]
  China | 90 | 89 | 179

OUTCOME MEASURES:

1. Primary Outcome: Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Cognition Domains
Description: The following 8 scales are combined into a single index that is normalized with a mean score of 100 and a standard deviation of 10. Higher scores are considered better cognitive performance. No subscales scores are reported and a final standardized score is reported as the average of the standardized scores on each of these scales. Here is the listing of component scales that were translated into Chinese and used for this study:
  Brief Assessment of Cognition in Schizophrenia (BACS): Symbol-Coding Trail Making Test: Part A Attention/Vigilance Continuous Performance Test-Identical Pairs (CPT-IP)* Wechsler Memory Scale®-3rd Ed. (WMS®-III): Spatial Span + Letter-Number Span Hopkins Verbal Learning Test-Revised™ (HVLT-R™) Brief Visuospatial Memory Test-Revised (BVMT-R™) Neuropsychological Assessment Battery® (NAB®): Mazes
  Mayer-Salovey-Caruso Emotional Intelligence Test (MSCEIT™):
Time Frame: end of 12 wk treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tropisetron | Placebo
Number analyzed (Participants) | 90 | 89
units on a scale | 96 (16) | 95 (15)
Statistical Analysis 1: Comparison: Tropisetron vs Placebo; Test type: Superiority or Other; p < 0.05, ANCOVA

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Tropisetron | Placebo
Serious Adverse Events (participants affected / at risk) | 0/90 | 0/89
Other Adverse Events (participants affected / at risk) | 8/90 | 6/89
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tropisetron (N=90) | Placebo (N=89)
Other Adverse Event (General disorders) | 8 (8) | 6 (6) — Dry mouth，Constipation, Blurred vision, Nausea

LIMITATIONS AND CAVEATS:
Since all participants were the first episode and drug naive patients, some participants quit before the completion of the entire clinical trial

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No